CLINICAL TRIAL: NCT01349647
Title: Immunization of Small Cell Lung Cancer Patients With a Pentavalent Vaccine Composed of KLH-conjugates of GD2L, GD3L, Globo H, Fucosyl GM1, and N-Propionylated Polysialic Acid
Brief Title: Immunization With a Pentavalent Vaccine Composed of KLH-conjugates of GD2L, GD3L, Globo H, Fucosyl GM1, and N-Propionylated Polysialic Acid
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-095
Record Dates: First submitted 2011-05-05; First posted 2011-05-06 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Lung Cancer
Keywords: FUCOSYL-GM1-KLH; GLOBO H-KLH CONJUGATE; OPT-821; POLYSIALIC ACID - KLH; Vaccine; 08-095
MeSH Terms: conditions — Lung Neoplasms | interventions — Globo-H; fucosyl GM1 ganglioside; Biological Products

ARMS (2):
- Vaccine and Chemotherapy (Experimental): This is a pilot trial evaluating the safety and immunogenicity of a pentavalent vaccine for patients with small cell lung cancer (SCLC). Patients with SCLC who have completed all planned initial therapy and have maintained a partial or complete response will be enrolled.
  Interventions: Biological: vaccine comprised of KLH conjugates of GD2L, GD3L, Globo H, fucosyl GM1, and N-propionylated polysialic acid plus OPT-821 adjuvant
- Vaccine Alone (Experimental): Patients will be vaccinated with the pentavalent vaccine comprised of KLH conjugates of GD2L, GD3L, Globo H, fucosyl GM1, and N-propionylated polysialic acid plus OPT-821 adjuvant.
  Interventions: Biological: Biological/Vaccine: vaccine comprised of KLH conjugates of GD2L, GD3L, Globo H, fucosyl GM1, and N-propionylated polysialic acid plus OPT-821 adjuvant

INTERVENTIONS:
Biological: vaccine comprised of KLH conjugates of GD2L, GD3L, Globo H, fucosyl GM1, and N-propionylated polysialic acid plus OPT-821 adjuvant — Patients will be vaccinated with the pentavalent vaccine comprised of KLH conjugates of GD2L, GD3L, Globo H, fucosyl GM1, and N-propionylated polysialic acid plus OPT-821 adjuvant. Patients will receive vaccine at weeks 1, 2, 3, 9, 20, and 32. Patients will also receive one cycle of chemotherapy with etoposide and cisplatin or carboplatin at week 6.
  Arms: Vaccine and Chemotherapy
Biological: Biological/Vaccine: vaccine comprised of KLH conjugates of GD2L, GD3L, Globo H, fucosyl GM1, and N-propionylated polysialic acid plus OPT-821 adjuvant — Patients will be vaccinated with the pentavalent vaccine comprised of KLH conjugates of GD2L, GD3L, Globo H, fucosyl GM1, and N-propionylated polysialic acid plus OPT-821 adjuvant.
  Patients will receive vaccine at weeks 1, 2, 3, 4, 8, and 16.
  Arms: Vaccine Alone

SUMMARY:
Even when small cell lung cancer responds well to treatment with chemotherapy, it has a tendency to grow back and to spread. The investigators are interested in testing new therapies aimed at decreasing this risk. This study tests a vaccine, which is a substance injected under the skin which can cause an immune response. The hope is that the body will make antibodies to the vaccine which will also react against the cancer. The vaccine is specific for small cell lung cancer. It combines several components (small cell lung cancer targets) that have been tested individually in patients with small cell lung cancer or other cancers (GD2, GD3, Globo H, Fucosyl GM1 and N-propionylated polysialic acid). Two other substances (KLH and OPT-821) are added which boost the immune system.

This study will have two groups of patients. The first group will receive the vaccines along with one cycle of chemotherapy. The second group will receive the vaccines without chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have small cell lung cancer confirmed by the Department of Pathology at Memorial Sloan-Kettering Cancer Center.
* Patients may have limited or extensive stage disease at the time of diagnosis.
* Patients must have completed first-line therapy, with or without thoracic and/or cranial irradiation, and have achieved either a complete response or partial response to therapy without subsequent evidence of disease progression.
* At least 3 weeks must have elapsed between the time the patient completed chemotherapy and the first vaccination.
* No more than 8 weeks can elapse between the time the patient completed chemotherapy and the first vaccination.
* If the patient received thoracic or cranial irradiation after completing the chemotherapy, at least 1 week must have elapsed after the radiation before the first vaccination. Patients must have recovered from the acute toxicities of the radiation prior to starting the vaccine therapy.
* Karnofsky Performance Status > or = to 70%.
* Hematologic parameters:
* WBC > or = to 3.0 x 10^3 cells/µl
* Total lymphocyte count > or = to 0.5 x 10^3 cells/µl
* Platelet count > 100,000/µl
* Biochemical parameters
* Creatinine clearance > or = to 40 ml/min
* Total bilirubin < or = to 1.5 x upper limits of normal
* AST and ALT < or = to 2.5 x upper limits of normal
* Patients must be able to give written informed consent.
* Patients must be ≥ 18 years old.

Exclusion Criteria:

* Patients with progression of disease after first-line chemotherapy.
* Pregnant or lactating women.
* Patients with a history of immunodeficiency or autoimmune disease, or who have undergone radiation to the spleen or splenectomy.
* Patients with a history of leptomeningeal disease.
* Patients with active infection requiring systemic antibiotics, antiviral, or antifungal treatments.
* Patients with serious unstable medical illness.
* Patients taking systemic corticosteroids.
* Patients with peripheral sensory neuropathy > grade 1.
* Patients who have used non-steroidal anti-inflammatory medications within 2 weeks of vaccination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Confirm the safety of the pentavalent vaccine in this patient population | 1 year
  After immunization with a pentavalent vaccine, including KLH conjugates of GD2L, GD3L, Globo H, fucosyl GM1, and N-propionylated polysialic acid, with the adjuvant OPT-821. Toxicity will be graded in accordance with Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. The vaccination will be considered safe if no more than 1 patient has new grade 2 neurotoxicity, grade 3 hepatotoxicity, new autoimmunity or grade 4 local or grade 3 systemic toxicity requiring cessation of treatment.
Confirm the immunogenicity of the pentavalent vaccine in this patient population | 1 year
  an antibody titer of > or = to 1:80 by ELISA against a given antigen or an ELISA titer > or = to 8 fold increase over baseline for patients with a detectable baseline titer; ) confirmation by FACS against tumor cells expressing the four antigens. An increase in percent positive cells by FACS by 3-fold (over 30%) compared to pretreatment level, with the pretreatment level set at 10%, is a positive FACS response.

SECONDARY OUTCOMES:
To measure the B-cell response at the cellular level | 1 year
  by generating and analyzing monoclonal antibodies against GD2L, GD3L, Globo H, Fucosyl GM1, and NPropionylated Polysialic Acid and to compare the avidity of the induced antigen specific IgG and IgM antibodies which is not possible with sera
To evaluate the use of a circulating tumor cell (CTC) assay in this patient population. | 1 year
  with minimal residual disease to determine if levels correlate with recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Krug, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm